CLINICAL TRIAL: NCT02045875
Title: Improving Asthma Control in the Real World: A Systematic Approach to Improving Dulera Adherence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asthma Management Systems (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); West Penn Allegheny Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC-5816
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-02

CONDITIONS: Asthma
Keywords: Adherence monitoring; Motivational Interviewing Adherence strategies
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate, Formoterol Fumarate Drug Combination; Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dulera adherence monitoring (Experimental): Adherence Monitoring Dulera; Identification of adherence barrier(s); Motivational Interviewing Adherence Strategies to promote adherence
  Interventions: Drug: Dulera
- Dulera Standard of Asthma Care (Active Comparator): Dulera standard of asthma care
  Interventions: Drug: Dulera

INTERVENTIONS:
Drug: Dulera — Dulera is a combination product containing a corticosteroid and a long-acting beta2-adrenergic agonist, FDA approved and indicated for treatment of asthma in patients 12 years of age and older.
  Other Names: mometasone furoate/formoterol fumarate dihydrate

SUMMARY:
40 subjects with moderate-to-severe asthma will be randomly selected for study in which 20, will be monitored for medication use (Dulera 100/5, Dulera 200/5 and Proventil HFA) over 3 months. These intervention subjects will receive medication use feedback at each visit, while the control group will receive the standard of asthma care. Those interventional subjects with Dulera adherence<60% will receive feedback based on an asthma adherence disease management model protocol, Asthma Adherence Pathway. Intervention clinicians will been trained in Motivational Interviewing to reduce subject ambivalence about medication use. The primary hypothesis is that subjects who receive medication monitoring and Motivational Interviewing adherence strategies will have better asthma control, as measured by the Asthma Control Questionnaire, than the control group.

DETAILED DESCRIPTION:
Primary Clinical Hypothesis: Poorly controlled subjects with moderate-to-severe asthma (measured by Asthma Control Questionnaire (ACQ) ≥ 1) despite treatment with Dulera, who are treated with the asthma adherence disease management protocol, Asthma Adherence Pathway™, will achieve greater asthma control than similar control subjects who are treated with the current standard of care.

Primary end point: There will be four measures of Asthma Control Questionnaire (ACQ) over time over 3 months. The primary endpoint is the third month measure of ACQ.

Secondary Clinical Hypothesis: The asthma adherence disease management program, Asthma Adherence Pathway™, will increase observed adherence to Dulera relative to a benchmark of 60% adherence (i.e., expected prescribed actuations).

Secondary end points: a) Average adherence to Dulera over the three month study period

Tertiary Clinical Hypothesis: Responses to Adult Asthma Adherence Questionnaire (AAAQ) will be related to Dulera Adherence

Tertiary Study Endpoints: There will be 2 measures of the AAAQ (first and last visit) and the tertiary endpoint is the last visit

ELIGIBILITY:
Inclusion Criteria:

1. Physician diagnosis of asthma of moderate severity
2. Subjects ≥ 18 years of age
3. Currently receiving an inhaled corticosteroid medication and being prescribed Dulera 100/5 as part of standard of care based upon asthma severity and dosing guidelines
4. Asthma Control Questionnaire (ACQ) result > 1.0 at entry
5. Demonstration of correct inhalation technique for use of meter-dosed inhalers (MDIs)
6. History of reversible airway obstruction documented by treating physician Exclusion Criteria: intermittent asthma; emphysema, chronic obstructive pulmonary disease; chronic bronchitis; cystic fibrosis; medication that may have a drug interaction with Dulera

Exclusion Criteria

1. Intermittent asthma (asthma exacerbations or symptoms < 3 days/week)
2. Diagnosis of emphysema in prior year
3. Diagnosis at any time of: chronic obstructive pulmonary disease (COPD), chronic bronchitis, cystic fibrosis, bronchiectasis, Churg Strauss, Wegener's, sarcoidosis, pulmonary hypertension or lung cancer
4. On any medication documented to have a drug interaction with Dulera

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03-04 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Gentile, DO, Principal Investigator — West Penn Allegheny Health System
Locations (1):
- West Penn Allegheny Health System, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dulera Adherence Monitoring | Dulera Standard of Asthma Care
Started | 27 | 23
Completed | 20 | 20
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dulera Adherence Monitoring | Dulera Standard of Asthma Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Full Range); unit: years] | 41 [23 to 67] | 39 [26 to 69] | 40 [23 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 8 | 5 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control
Description: Asthma Control Questionnaire measured at each office visit. ACQ integrates values by 6 clinical questions related to symptoms and the value related to FEV1% predicted with a total score ranging from 0-6 and higher values indicating poorer asthma control.
Time Frame: Baseline, one, two and three months
Population: All patients who completed ACQ at 4 clinical visits were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dulera Adherence Monitoring | Dulera Standard of Asthma Care
Number analyzed (Participants) | 19 | 20
units on a scale
  baseline | 1.857 (0.924) | 1.592 (0.839)
  one month | 1.792 (1.359) | 1.578 (0.855)
  two month | 1.345 (1.184) | 1.488 (0.947)
  three month | 1.105 (0.806) | 1.407 (0.759)
Statistical Analysis 1: Comparison: Dulera Adherence Monitoring vs Dulera Standard of Asthma Care; Test type: Superiority; p = 0.046, ANOVA — Effect of interaction of time and treatment group

2. Secondary Outcome: Adherence to Dulera 100/5 and 200/5
Description: Subjects in the monitoring group will have adherence greater than or equal to the 60% benchmark
  Adherence was calculated by taking the number of doses actually taken divided by the number of doses prescribed and multiplying by 100.
Time Frame: week 2. months 1, 2, and 3
Population: Data was only collected in the interventional group.
Measure: Mean (Standard Deviation); unit: percent of prescribed doses
Arm/Group | Dulera Adherence Monitoring
Number analyzed (Participants) | 20
percent of prescribed doses
  week 2 | 88.75 (10.43)
  month 1 | 80.7 (14.52)
  month 2 | 77.55 (19.13)
  month 3 | 76.8 (19.83)
Statistical Analysis 1: Comparison: Dulera Adherence Monitoring; Test type: Other; correlation coefficient = -0.508 — correlation of asthma control and adherence

3. Secondary Outcome: Overall Adherence to Dulera 100/5 and 200/5
Description: Subjects in the monitoring group will have adherence greater than or equal to the 60% benchmark
  Overall interval value was the mean of daily percent
Time Frame: 3 months
Population: Data was only collected in the interventional group.
Measure: Mean (Standard Deviation); unit: percent of prescribed doses per day
Arm/Group | Dulera Adherence Monitoring
Number analyzed (Participants) | 20
percent of prescribed doses per day | 80.95 (14.23)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Dulera Adherence Monitoring | Dulera Standard of Asthma Care
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/23
Other Adverse Events (participants affected / at risk) | 0/27 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT02045875/Prot_SAP_000.pdf